CLINICAL TRIAL: NCT06033066
Title: A Randomized Trial of Financial Incentives for the Recruitment of County Health System Patients to the Alzheimer Prevention Trials (APT) Webstudy
Brief Title: Financial Incentives and Recruitment to the APT Webstudy
Acronym: FIND-AD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: American Heart Association (Other); Schaeffer Center for Health Policy & Economics (Unknown); Alzheimer's Therapeutic Research Institute (Other)
Responsible Party: Principal Investigator, Mireille Jacobson, Associate Professor of Gerontology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UP-22-01037
Record Dates: First submitted 2023-08-09; First posted 2023-09-13 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease; Dementia; Preclinical Alzheimer's Disease; Prodromal Alzheimer's Disease
Keywords: Alzheimer's; Prevention; Observational; Trial-Ready Cohort
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Messaging Only (Active Comparator): 16,000 participants will be randomized to Arm 1 where no monetary incentive is offered.
  Interventions: Behavioral: Message
- Small Incentive (Experimental): 16,000 participants will be randomized to Arm 2 where a small one-time monetary incentive is offered.
  Interventions: Behavioral: Financial Incentives
- Prize Incentive (Experimental): 16,000 participants will be randomized to Arm 3 where an opportunity based incentive (or a drawing with a prize) with a single winner will be offered.
  Interventions: Behavioral: Financial Incentives

INTERVENTIONS:
Behavioral: Financial Incentives — Small financial incentive or prize incentive
  Arms: Prize Incentive; Small Incentive
Behavioral: Message — Message inviting participant to enroll
  Arms: Messaging Only

SUMMARY:
This single-blind, three-arm, randomized, controlled trial will assess the impact of messages and financial incentives on the enrollment of demographically diverse individuals to the Alzheimer Prevention Trials (APT) Webstudy. The APT Webstudy is a novel, online registry that employs quarterly cognitive testing using validated platforms. The APT Webstudy implements fully remote assessments, coordinated by the Alzheimer's Therapeutic Research Institute (ATRI) under USC IRB #HS-17-00746. The purpose of the current study is to test whether we can increase enrollment of diverse individuals into the registry. To do this, we will work with Contra Costa Regional Medical Center (CCRMC), the county public hospital and its affiliated health centers in Contra Costa County, California, to test whether sending messages with and without financial incentives to patients who receive primary care with the health system can increase enrollment to the APT Webstudy. The investigators hypothesize that 1) a certain small financial incentive and an award opportunity based incentive (or a drawing with a prize) will increase enrollment rates of CCHS members into the APT Webstudy relative to the control group. The investigators further hypothesize that the award opportunity incentive will increase the enrollment rate of CCRMC patients into the APT Webstudy more than a certain financial incentive with the same expected value.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all of the following criteria:

* Patients empaneled at Contra Costa Regional Medical Center (CCRMC), the county public hospital and its affiliated health centers.
* Age 50 or older
* Literate in either English or Spanish

Exclusion Criteria:

* Below age 50
* Documentation of prior dementia diagnosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44844 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Enrollment status into the APT Webstudy | 2-weeks
  APT Webstudy enrollment rate based on completion of at least one of the two APT Webstudy cognitive assessments (Cognitive Function Instrument [CFI] and/or Cogstate Brief Battery).

SECONDARY OUTCOMES:
Cost per enrollee | annual
  Cost to acquire an enrollment
Completion of cognitive assessments within the APT Webstudy | 2-weeks
  Completion of both APT Webstudy cognitive assessments (Cognitive Function Instrument [CFI] and/or Cogstate Brief Battery).

CONTACTS AND LOCATIONS:
Locations (1):
- Contra Costa Health Plan, Martinez, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The health system will not allow sharing of individual data on a public site. However, we will share data on request from investigators.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available within 6 months of publication.
Access Criteria: Individual data shared upon request.

REFERENCES:
- [Derived] Jacobson M, Molina-Henry D, Chang TY, Jimenez-Maggiora GA, Pramanik R, Shah SB, Aisen PS. Financial Incentives to Increase Diversity of Older Participants in a Memory Concerns Registry: A Randomized Clinical Trial. JAMA Health Forum. 2025 Aug 1;6(8):e252273. doi: 10.1001/jamahealthforum.2025.2273. PMID 40844772
- See also: APT Webstudy — https://www.aptwebstudy.org/

DOCUMENTS (1):
  • Study Protocol (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT06033066/Prot_000.pdf